CLINICAL TRIAL: NCT00579072
Title: The Impact of Androgen Ablation Therapy on Cognitive Functioning and Functional Status in Men With Prostate Cancer Age 65 and Older
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); City of Hope National Medical Center (Other); Fordham University (Other); Columbia University (Other); NYU Langone Health (Other); Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 06-084
Record Dates: First submitted 2007-12-19; First posted 2007-12-21 (Estimated); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer
Keywords: Prostate; cognitive effects; 06-084
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Longitudinal Study: Take part in this study because subject has prostate cancer and are over 64 years old. To run this study,need men from two groups. First, we need men who are about to start hormone treatment. Second, we need men who do not plan to use this treatment in the future. We will use this second group as a control group and compare this group to the men who are using this treatment.
  Interventions: Behavioral: Questionaires; Device: fMRI scan (optional)
- Group Comparison: Take part in this study because subject has prostate cancer and are over 64 years old. Also, because subject has been on hormone therapy for about two to three years.
  Interventions: Behavioral: Questionaires; Device: fMRI scan (optional)

INTERVENTIONS:
Behavioral: Questionaires — We will use a 6-month longitudinal design to assess the short-term cognitive effects of androgen ablation therapy. We will collect 6-month longitudinal data on 170 men with prostate cancer. All 170 men will be hormone naïve at the start of this study (Hormone Naïve Group). These 170 men will consist of two subgroups. The first subgroup will comprise 70 men with prostate cancer age 65 and older scheduled to start androgen ablation therapy. Their cognitive functioning will be assessed prior to starting androgen ablation therapy or within 21 days after initiation, (i.e. baseline) and then 6 months later (Androgen Ablation Subgroup).The second subgroup will serve as a control group, and consist of 100 men with prostate cancer age 65 and older who are at least 1-year post definitive localized treatment with no evidence of disease and no plan to start androgen ablation therapy (No Androgen Ablation Subgroup).
  Groups: Longitudinal Study
Behavioral: Questionaires — To supplement the pilot data collected in Aim 1, Aim 2 we will utilize a group comparison design to assess the long-term cognitive effects of androgen ablation therapy. We will collect data on the cognitive functioning of 110 men with prostate cancer age 65 and older who have been on continuous androgen ablation therapy for 1-3 years (2-Year Androgen Ablation Group). These men will complete the study battery once (i.e., the neuropsychological battery, psychosocial questionnaires, and a functional status battery). We will compare the cognitive functioning of these 110 men in the 2-Year Androgen Ablation Group to the 170 men with prostate cancer who are hormone naïve (Hormone Naïve Group).
  Groups: Group Comparison
Device: fMRI scan (optional) — Main study participants will be offered to complete an optional fMRI. Fifteen participants from the No Androgen Ablation Subgroup and 15 participants from the Comparison Androgen Ablation Subgroup or Longitudinal Androgen Ablation Subgroup will be recruited for this portion of the study. The fMRI will be scheduled either the same day as the neurocognitive assessment or within eight weeks of the neurocognitive testing. The fMRI will be performed only once at baseline for the Comparison Androgen Ablation Subgroup. The fMRI will be performed at the follow-up time point for the Longitudinal Androgen Ablation Subgroup. The fMRI will be performed at baseline for the No Androgen Ablation Subgroup; if the fMRI can not be completed at baseline (due to participant schedule conflict, lack of fMRI availability, staff schedule conflict, etc.), then the scan will be conducted at the follow-up time point if possible.

SUMMARY:
The purpose of this study is to find out if therapy with hormones (such as Lupron, Casodex, Zolodex or Degarelix) change a person's thinking abilities.

DETAILED DESCRIPTION:
To find out if this treatment changes things like memory, learning, or concentration. This study is being done to learn more about the effects of this treatment and to help men in the future who use the hormones Lupron, Casodex, Zolodex or Degarelix.

If you choose to take part, you will be asked to do the following:

Fill out questionnaires that ask about:

* Your age, eduction, race, and income
* Depression
* Stress
* Energy level
* Pain
* Memory
* Ability to perform daily tasks such as eating, dressing, and taking a shower

Research staff will evaluate you on the following:

* Memory
* How you prefer to learn new information
* Copying designs such as rectangles, squares, and circles
* How quickly you think
* Your attention span
* How well you plan and organize shapes and colors into specific categories

As such, at MSKCC will be contacting a portion of prospective subjects via mail or email to offer them the opportunity to plan for and allocate the necessary time in their personal schedules, should they be interested in the study.

ELIGIBILITY:
Inclusion Criteria is the same at both sites, and is outlined below:

Inclusion Criteria:

Comparison Androgen Ablation Group

1. Diagnosis of prostate cancer
2. Age 65 or older
3. Ability to converse, write and read English
4. In the investigator's judgment, participants must have satisfactory cognitive function to provide valid informed consent and participate in the neurocognitive testing. The Blessed Orientation-Memory-Concentration test (BOMC) will be used as a cognitive screening tool. Patients must have a BOMC score of less than or equal to 11.
5. Able to provide informed consent
6. Have been on continuous androgen ablation therapy for 6 months to-3 years

Longitudinal Androgen Ablation Subgroup

1. Diagnosis of prostate cancer
2. Age 65 or older
3. Ability to converse, write and read English
4. Able to provide informed consent
5. In the investigator's judgment, participants must have satisfactory cognitive function to provide valid informed consent and participate in the neurocognitive testing. The Blessed Orientation-Memory-Concentration test (BOMC) will be used as a cognitive screening tool. Patients must have a BOMC score of less than or equal to 11.
6. Starting androgen ablation therapy or started within the past 21 days
7. No androgen ablation therapy within the past year

No Androgen Ablation Subgroup

1. Diagnosis of prostate cancer
2. Age 65 or older
3. In the investigator's judgment, participants must have satisfactory cognitive function to provide valid informed consent and participate in the neurocognitive testing. The Blessed Orientation-Memory-Concentration test (BOMC) will be used as a cognitive screening tool. Patients must have a BOMC score of less than or equal to 11.
4. At least 1-year post definitive localized treatment
5. Ability to converse, write and read English
6. Able to provide informed consent
7. Not anticipated to start androgen ablation therapy
8. No history of androgen ablation therapy

Exclusion Criteria:

All Groups

1. Previous or current treatment with chemotherapy
2. As per medical record or self-report, a history of central nervous system stroke, history of traumatic brain injury, or diagnosis of neurogenerative disorder that affects cognitive function (e.g. Alzheimer's, Parkinson's, Multiple Sclerosis, dementia, seizure disorders, etc.)
3. History of untreated psychiatric disease
4. As per medical record or self-report, history of loss of consciousness for 60+ minutes and/or admitted to the hospital for a head injury
5. Current use of opioids
6. History of developmental disorders
7. Current or history of alcohol or substance abuse
8. Visual, auditory, or other impairment that would preclude ability to complete neuropsychological testing (e.g. significant macular degeneration, being unable to correct hearing with hearing aides, hand tremors, etc.)

CRITERIA FOR OPTIONAL fMRI

Exclusion Criteria:

* Patient has a self-reported fear of enclosed spaces (Claustrophobia)
* As per self report or as identified in the medical record, patient has any of the following items that preclude fMRI evaluation:
* Cardiac pacemaker
* Joint replacements
* Aneurysm clips
* Transdermal patched
* Aortic clips
* Prosthesis
* Intracranial bypass clips
* Harrington rod
* Coronary Artery bypass clips
* Biostimulator
* Renal Transplant Clips
* Bone or joint pins
* Other vascular clips or filters
* Tissue expander
* Implanted neurostimulators
* Metal mesh
* Artificial heart valve
* Stents
* Insulin pump
* Wire structures
* Electrodes
* Shrapnel/bullets
* Hearing Aids /implant
* Implanted electrical devices
* IUD Metal in eyes
* Shunts
* Ocular Implants
* Hair extensions
* Hair implants
* Tattoos above the waist
* Any possible metal in body
* As per self report, patient has dentures, body jewelry or wig that they are unable to remove

Min Age: 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Prostate Cancer Patients
Sampling Method: Non-Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2006-08; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Describe changes in cognitive functioning over 6 mos in 70 men with prostate cancer who are about to start androgen ablation therapy vs 70 men with prostate cancer with NED & no medical indication to start Comparison androgen ablation therapy | 3 years

SECONDARY OUTCOMES:
Describe differences in cognitive functioning in 80 men with prostate cancer who received Comparison androgen ablation therapy for 6 months - 3 years vs.140 men with prostate cancer who are hormone naïve. | 3 years
To describe the differences in cognitive functioning in 70 men with prostate cancer who have received androgen ablation therapy for 6 months vs. 80 men with prostate cancer who have received Comparison androgen ablation therapy for 6 months-3 years. | 3 years
To investigate regionally specific differences in brain activity mediated by testosterone. | 3 years
To investigate differences in neuropsychological performance on the mental rotation task and their relation to regional brain recruitment as demonstrated in the above outcome | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Christian Nelson, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - City of Hope, Duarte, California
  - Memorial Sloan Kettering Cancer Center, New York, New York

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm